CLINICAL TRIAL: NCT03838224
Title: Effects of a Single Dry Needling Session of the Obliquus Capitis Inferior on the Altered Sensorimotor Function in People With Neck Pain: a Random Control Trial
Brief Title: A Single Dry Needling Session of the Obliquus Capitis Inferior for the Altered Sensorimotor Function in People With Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Enrique Lluch Girbés, Principal investigator, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H1542206264486
Record Dates: First submitted 2019-01-29; First posted 2019-02-12 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Whiplash Syndrome; Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (Experimental): Participants allocated in this group will receive a single session of dry needling of the obliquus capitis inferior. Prior to the intervention, participants will receive information about the procedure and will be free to withdraw. The needle was shown to the participant before the intervention. Participants will be requested to lie in prone on the plinth. Participants' skin will be sterilized with antiseptic spray for the skin. The therapist will clean his hands and use sterilized gloves.
  Interventions: Other: dry needling
- sham needling (Sham Comparator): Sham needling has shown to be a valid control method in dry needling research. The procedure in the sham group will be the same as the experimental group to guarantee the participants' blinding. Prior to the intervention, participants will receive information about the procedure and will be free to withdraw. The sham needle (same appearance/material as the true needle) was shown to the participant before the intervention to guarantee the blinding.
  Interventions: Other: Sham needling

INTERVENTIONS:
Other: dry needling — Participants allocated in this group will receive a single session of dry needling of the obliquus capitis inferior. Prior to the intervention, participants will receive information about the procedure and will be free to withdraw. The needle was shown to the participant before the intervention. Participants will be requested to lie in prone on the plinth. Participants' skin will be sterilized with antiseptic spray for the skin. The therapist will clean his hands and use sterilized gloves. The needle will be moved up and down within the muscle, using a "fast-in and fast-out" technique. Needle insertions will be repeated 12 times.
  Arms: Dry needling
Other: Sham needling — Sham needling has shown to be a valid control method in dry needling research. The procedure in the sham group will be the same as the experimental group to guarantee the participants' blinding. Prior to the intervention, participants will receive information about the procedure and will be free to withdraw. The sham needle (same appearance/material as the true needle) was shown to the participant before the intervention to guarantee the blinding.
  Arms: sham needling

SUMMARY:
Neck pain is the 3rd cause of disability worldwide and represents an enormous socioeconomic burden. It has been reported that people with neck pain, with traumatic and non-traumatic onset, have an alteration of the sensorimotor function compared to pain-free people, such as deficits in the head and neck repositioning or alteration of the body balance. It has been suggested that alterations on the proprioception of the suboccipital muscles may cause a decrease in head and neck repositioning accuracy and changes in head and neck positioning patterns. The suboccipital muscles, particularly the obliquus capitis inferior (OCI), has a greater density of muscular spindles compared to lower cervical segments, which is believed to play an important role in the proprioception. The alteration of the JPE is more often found in patients with a dysfunction in the upper cervical spine, but people with lower dysfunction can also exhibit it. However, no conclusive results on JPE have been reported with articular techniques targeting the upper cervical spine. On the contrary, positive results on this test have been observed after the retraining of the upper cervical muscles. As OCI is a deep muscle, dry needling seems to be the most appropriate passive modality of treatment to target that muscle and restore the abnormal cervical sensorimotor control. However, this hypothesis has never been tested.

DETAILED DESCRIPTION:
The aim of the proposed study is to investigate if a single dry needling (DN) session modifies the altered sensorimotor function in people with neck pain. The secondary objectives will be to investigate the effects of a single DN session on muscle length (indirectly measured with FRT) and to investigate the effects of a single DN session on self-reported pain.

With this aim, a random control trial (RCT) design will be conducted with two groups; intervention group (dry needling of the OCI) and placebo group (sham needling). Sham needling has shown to be a valid control method in dry needling research.

The study will take two days. In the first day, the outcome measures will be measured before (baseline) and immediately after the intervention (immediate follow-up). In the second day (one-week follow-up), outcome measures will be measured again. Pain intensity, measured with the visual analogue scale, will be only measured at baseline and one-week follow-up.

The baseline and follow-up assessments will be performed by an independent assessor who will be blinded to the intervention allocation. The interventions will be provided by a therapist with dry needling training and 3-years of musculoskeletal experience who will be blinded to outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Neck pain longer than 3 months (traumatic or non-traumatic)
* Neck disability index (NDI) ≥10
* Visual analogue scale (VAS) ≥3
* Joint position error (JPE) ≥4.5º determined in the physical examination prior to enrollment

Exclusion Criteria:

* Previous cervical spine surgery
* Spine fracture
* Any neurological signs
* Cervical stenosis
* Needle phobia/fear of needles
* Anticoagulant medication consumption
* Pregnancy
* Known or suspected vestibular pathology
* Vertigo or dizziness from ear or brain disorders, sensory nerve pathways (e.g. BPPV).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Joint position error (JPE) | Baseline, immediate post-intervention follow-up and one-week post-intervention follow-up
  Cervical JPE will be measured using a laser-pointer attached to a lightweight headband. In sitting position, 90 cm away from a target and blindfolded, patients will be requested to rotate to the right and to the left. An absolute error between the starting and end points will be calculated in millimeters and then converted to degrees. Six repetitions will be performed each side according to recommendations and the mean will be calculated.

SECONDARY OUTCOMES:
Change in Cervical movement sense | Baseline, immediate post-intervention follow-up and one-week post-intervention follow-up
  Participants will trace with the laser-pointer in their heads a specific pattern (located at 100 cm distance) at two velocities (accurate; accurate and fast). This test will be recorded and later examined at slow motion by a video analysis programme. Time (total time taken to complete the pattern), error frequency (number of deviations) and error magnitude (sum of deviations multiplied by the distance from the central line) will be measured. This test has shown high intra and inter-rater reliability.
Change in Postural stability | Baseline, immediate post-intervention follow-up and one-week post-intervention follow-up
  Patients will be positioned on the force platform. The postural sway will be measured in 4 conditions as follows: (neutral) narrow stance (feet close together) on firm and soft surfaces with eyes open and eyes closed
Change in Active cervical range of motion (rotation) | Baseline, immediate post-intervention follow-up and one-week post-intervention follow-up
  Cervical ROM in rotation will be measured bilaterally with the patients in sitting position using a Cervical Range of Motion (CROM) instrument, which has been shown to be a reliable and valid tool.
Change in Cervical flexion-rotation test (CFRT) | Baseline, immediate post-intervention follow-up and one-week post-intervention follow-up
  Upper cervical ROM in rotation will be measured bilaterally with the CFRT using the CROM. Participants will be requested to lie in supine on the plitch and the examiner will perform rotation passively with the rest of the cervical spine blocked in full flexion position. This test has shown to be a valid and reliable tool to measure the range of motion of the upper cervical spine (C1-C2).
Change in Smooth pursuit neck torsion (SPNT) | Baseline, immediate post-intervention follow-up and one-week post-intervention follow-up
  This test is understood to assess eye movement disturbances due to altered cervical afferent input. Patients will be sat in a neutral position on a swivel chair and will be requested to follow a pen in the hand of the examiner (with their eyes) whilst keeping their head still. The pen will be moved at the participant's natural focal length across their field of vision horizontally in a visual range of 40 degrees several times. The speed of the movement will be 20 degrees per second. Pursuit of the eyes will be observed. The test will be repeated with the neck torsioned to the left and right by rotating the trunk and shoulders to the right 45 degrees, keeping the head still. This is done so that input to the vestibular system is avoided.
  Increased catch up saccades in the torsion position especially as they cross the midline and/or reproduction of symptoms in the torsion position compared to the neutral position is a positive test.
Change in Neck pain intensity | Baseline and one-week post-intervention follow-up
  Neck pain intensity will be measured using a visual analogue scale (VAS). Patients will be requested to grade their pain intensity of neck pain experienced on a 0-100 mm horizontal line (0 mm= no pain and 100 mm= worst pain imaginable).

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Lluch, PhD, Study Director — Physiotherapy Department University of Valencia
Locations (1):
- University of Valencia, Valencia, Spain

REFERENCES:
- [Background] Jull G, Falla D, Treleaven J, Hodges P, Vicenzino B. Retraining cervical joint position sense: the effect of two exercise regimes. J Orthop Res. 2007 Mar;25(3):404-12. doi: 10.1002/jor.20220. PMID 17143898
- [Background] Kulkarni V, Chandy MJ, Babu KS. Quantitative study of muscle spindles in suboccipital muscles of human foetuses. Neurol India. 2001 Dec;49(4):355-9. PMID 11799407
- [Background] Mitchell UH, Stoneman P, Larson RE, Page GL. The Construction of Sham Dry Needles and Their Validity. Evid Based Complement Alternat Med. 2018 Jun 14;2018:9567061. doi: 10.1155/2018/9567061. eCollection 2018. PMID 30013605
- [Background] Reid SA, Callister R, Katekar MG, Rivett DA. Effects of cervical spine manual therapy on range of motion, head repositioning, and balance in participants with cervicogenic dizziness: a randomized controlled trial. Arch Phys Med Rehabil. 2014 Sep;95(9):1603-12. doi: 10.1016/j.apmr.2014.04.009. Epub 2014 May 2. PMID 24792139
- [Background] Revel M, Andre-Deshays C, Minguet M. Cervicocephalic kinesthetic sensibility in patients with cervical pain. Arch Phys Med Rehabil. 1991 Apr;72(5):288-91. PMID 2009044
- [Background] Treleaven J, Clamaron-Cheers C, Jull G. Does the region of pain influence the presence of sensorimotor disturbances in neck pain disorders? Man Ther. 2011 Dec;16(6):636-40. doi: 10.1016/j.math.2011.07.008. Epub 2011 Sep 3. PMID 21890397
- [Background] Hallgren RC, Andary MT, Wyman AJ, Rowan JJ. A standardized protocol for needle placement in suboccipital muscles. Clin Anat. 2008 Sep;21(6):501-8. doi: 10.1002/ca.20660. PMID 18627103
- [Background] Audette I, Dumas JP, Cote JN, De Serres SJ. Validity and between-day reliability of the cervical range of motion (CROM) device. J Orthop Sports Phys Ther. 2010 May;40(5):318-23. doi: 10.2519/jospt.2010.3180. PMID 20436238
- [Background] Hall T, Robinson K. The flexion-rotation test and active cervical mobility--a comparative measurement study in cervicogenic headache. Man Ther. 2004 Nov;9(4):197-202. doi: 10.1016/j.math.2004.04.004. PMID 15522644
- [Background] Hall TM, Robinson KW, Fujinawa O, Akasaka K, Pyne EA. Intertester reliability and diagnostic validity of the cervical flexion-rotation test. J Manipulative Physiol Ther. 2008 May;31(4):293-300. doi: 10.1016/j.jmpt.2008.03.012. PMID 18486750
- [Background] Kamper SJ, Grootjans SJ, Michaleff ZA, Maher CG, McAuley JH, Sterling M. Measuring pain intensity in patients with neck pain: does it matter how you do it? Pain Pract. 2015 Feb;15(2):159-67. doi: 10.1111/papr.12169. Epub 2014 Jan 17. PMID 24433369
- [Background] Silva AG, Cruz AL. Standing balance in patients with whiplash-associated neck pain and idiopathic neck pain when compared with asymptomatic participants: A systematic review. Physiother Theory Pract. 2013 Jan;29(1):1-18. doi: 10.3109/09593985.2012.677111. Epub 2012 Apr 20. PMID 22515180
- [Background] Swait G, Rushton AB, Miall RC, Newell D. Evaluation of cervical proprioceptive function: optimizing protocols and comparison between tests in normal subjects. Spine (Phila Pa 1976). 2007 Nov 15;32(24):E692-701. doi: 10.1097/BRS.0b013e31815a5a1b. PMID 18007229
- [Background] Takasaki H, Hall T, Oshiro S, Kaneko S, Ikemoto Y, Jull G. Normal kinematics of the upper cervical spine during the Flexion-Rotation Test - In vivo measurements using magnetic resonance imaging. Man Ther. 2011 Apr;16(2):167-71. doi: 10.1016/j.math.2010.10.002. Epub 2010 Nov 4. PMID 21055995
- [Background] Werner IM, Ernst MJ, Treleaven J, Crawford RJ. Intra and interrater reliability and clinical feasibility of a simple measure of cervical movement sense in patients with neck pain. BMC Musculoskelet Disord. 2018 Oct 5;19(1):358. doi: 10.1186/s12891-018-2287-0. PMID 30290759